CLINICAL TRIAL: NCT03827967
Title: A Phase Ib Trial of Neoadjuvant PalloV-CC (Particle-delivered, Allogeneic Tumor Cell Lysate Vaccine for Colon Cancer) in Colon Cancer
Brief Title: Trial of PalloV-CC in Colon Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: George E. Peoples (Industry)
Responsible Party: Sponsor-Investigator, George E. Peoples, CEO, Cancer Insight, LLC, Cancer Insight, LLC
Organization: Cancer Insight, LLC (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PV-CC-01
Record Dates: First submitted 2018-09-11; First posted 2019-02-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Treatment cohorts (each n=6 total of n=24):
  1. 1 x 10^8 particles of PalloV-CC
  2. 2 x 10^8 particles of PalloV-CC
  3. 4 x 10^8 particles of PalloV-CC
  4. 8 x 10^8 particles of PalloV-CC PalloV-CC is inoculated weekly via intradermal injection. There will be sequential enrollment of dose-escalation cohorts, each patient treatment period is 4 weeks. Patients will conclude treatment with colectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1x10^8 particles of PalloV-CC (Experimental): Intradermal injection of PalloV-CC weekly x 4 weekly
  Interventions: Biological: PalloV-CC
- 2x10^8 particles of PalloV-CC (Experimental): Intradermal injection of PalloV-CC weekly x 4 weekly
  Interventions: Biological: PalloV-CC
- 4x10^8 particles of PalloV-CC (Experimental): Intradermal injection of PalloV-CC weekly x 4 weekly
  Interventions: Biological: PalloV-CC
- 8x10^8 particles of PalloV-CC (Experimental): Intradermal injection of PalloV-CC weekly x 4 weekly
  Interventions: Biological: PalloV-CC

INTERVENTIONS:
Biological: PalloV-CC — The PalloV-CC vaccine uses yeast cell wall particles (YCWP) to serve as an efficient vaccine delivery system as they can contain a broad range of antigenic material, they are rapidly phagocytized by antigen presenting cells, and they are inherently immunogenic. The PalloV-CC vaccine utilizes silicate-capped YCWP to deliver allogenic colon cancer tumor lysate. The vaccine will be given to subjects with resectable colon cancers neoadjuvantly shortly before surgery in order to study the effect of the vaccine on the tumor microenvironment using a well-validated immune scoring system for colon cancer and other immunologic tests.

SUMMARY:
This study is a phase Ib prospective, open label study evaluating the effect of vaccination on the immune microenvironment of cancers with results compared to banked tissue from historical controls. Prospectively vaccinated patients will also serve as their own controls by comparing the immune microenvironment of the tumor in pre-treatment biopsies to post-treatment surgical specimens. This is also a dose-escalation study with consecutive enrollment and advancement of cohorts in an overlapping fashion.

DETAILED DESCRIPTION:
This is a single arm, open label, phase Ib trial of neoadjuvant vaccination in colon cancer. The primary endpoint is the safety and toxicity of the vaccine. The primary immunologic endpoint is the impact of vaccination on the tumor microenvironment compared to prospectively evaluated, tissue banked specimens from historical controls. The tumor microenvironment will also be compared in matched pre- and post-treatment tissue samples in vaccinated subjects. Patients with endoscopic biopsy proven colon cancer will be identified by the staff in the gastroenterology, surgery, and/or the hematology/oncology clinics at the individual study sites. A research nurse, study coordinator, or study investigator will approach these patients about being in the trial and will introduce the trial to the prospective volunteer patient. If the patient is interested and appears eligible, the nurse, study coordinator, or investigator will arrange an appointment to counsel and consent the patient. Once consent is obtained, the nurse, study coordinator, or investigator will thoroughly screen the patient for inclusion and exclusion eligibility criteria.

If volunteers meet all inclusion criteria and none of the exclusion criteria and agree to participate, they will continue in the study, consented and enrolled for treatment assignment. Enrollment will start in cohort 1 with enrollment of 6 patients, and follow sequentially into the remaining cohorts, until all cohorts are completed. After treatment of all 6 patients in each dose cohort, a comprehensive safety analysis will be performed for short-term toxicity. If no dose limiting toxicity (DLT, >grade 2, related, or serious adverse event (SAE)) is found, then the next cohort will be enrolled. If three patients in a given dose cohort experience a DLT, then that dose will be determined to be the maximal tolerated dose (MTD), and the next dose cohort will not be initiated. At the completion of dosing of cohorts (last surgical colectomy performed), a comprehensive safety analysis will be performed for long-term toxicity. If the MTD is not reached, then a total of 24 patients will be enrolled.

Treatment cohorts (each n=6, total of n=24):

1. 1 x 10^8 particles of PalloV-CC
2. 2 x 10^8 particles of PalloV-CC
3. 4 x 10^8 particles of PalloV-CC
4. 8 x 10^8 particles of PalloV-CC

PalloV-CC is inoculated weekly via intradermal injection. There will be sequential enrollment of dose-escalation cohorts (Appendix A), each patient treatment period is 4 weeks (Appendix B). Patients will conclude treatment with colectomy.

Safety data will be collected on local and systemic toxicities and graded and reported per the Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

A total of 190 mL of blood will be drawn throughout the course of the study over a 3-4 week period. The patient will have 70mL of blood drawn for the following: a CBC with differential (10 mL of blood), a CMP (10 mL of blood), and study blood (50 mL of blood). This will be drawn on two separate occasions: once prior to the first vaccine inoculation, and again after the completion of the final vaccine inoculation (but prior to surgery). An additional 50 mL of study blood will be drawn midway through the vaccine series (at the third inoculation).

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-IV (resectable) colon cancer patients identified prior to their definitive surgery
2. Diagnosis definitively confirmed by endoscopic biopsy with tumor tissue slides available for analysis
3. Asymptomatic and capable of waiting 4 weeks prior to definitive surgery
4. ECOG 0-1 performance
5. Not involved in other clinical trials
6. Capable of giving informed consent

Exclusion Criteria:

1. Symptoms of obstruction or GI bleeding that necessitate more urgent surgical intervention
2. Cancer not definitively confirmed on endoscopic biopsy (i.e., Only high-grade dysplasia or adenoma identified, even if malignancy is suspected)
3. Known immune deficiency disease or HIV, active HBV, or active HCV
4. Steroids or other immunosuppressants received within 6 weeks of enrollment
5. Any colon cancer directed treatment (chemotherapy or radiation) received or planned prior to surgical resection
6. A history of any hematologic malignancy or myeloproliferative disease within 5 years prior to enrollment
7. Leukopenia or neutropenia within two weeks of presentation
8. ECOG >/= 2
9. Pregnancy (serum or urine HCG) or breast feeding
10. Tbili >1.8, Cr >2, Hgb <10, platelet count <50,000, WBC <2,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint-Overall number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 1 year for all 4 cohorts to enroll and undergo treatment.
  To determine the overall safety and toxicity of the PalloV CC vaccine by analyzing number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Primary Safety Endpoint-Per Dosing Cohort number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 1 year for all 4 cohorts to enroll and undergo treatment.
  To determine the safety and toxicity of the PalloV CC vaccine per dosing cohorts by analyzing number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Primary Immunologic Endpoint-Overall Immunoscore of the tumor microenvironment | 1 year for all 4 cohorts to enroll and undergo treatment.
  To determine the effect of vaccination on the tumor microenvironment in colon cancer by comparing the proportion of subjects with high Immunoscore (scale range: low, intermediate, high) in all vaccinated subjects to historical control subjects.
Primary Immunologic Endpoint-Per Dosing Cohort Immunoscore of the tumor microenvironment | 1 year for all 4 cohorts to enroll and undergo treatment.
  To determine the effect of vaccination on the tumor microenvironment in colon cancer by comparing the proportion of subjects Immunoscore (scale range: low, intermediate, high) in vaccinated subjects per dosing cohorts to historical control subjects Immunoscore (scale range: low, intermediate, high).

SECONDARY OUTCOMES:
Secondary Endpoint-Effect Tumor Microenvironment measured via Immunoscore | 1 year for all 4 cohorts to enroll and undergo treatment.
  To determine the effect of vaccination on the tumor microenvironment in colon cancer by comparing the Immunoscore (scale range: low, intermediate, high) between matched endoscopic biopsies (pre-vaccination) and resected final specimens (post-vaccination).
Secondary Endpoint-Immunologic comparison of evaluations of tumor microenvironment | 1 year for all 4 cohorts to enroll and undergo treatment.
  To determine the concordance of Immunoscore (scale range: low, intermediate, high) with other emerging analytical tools such as gene expression data analysis (CIBERSORT) and T-cell receptor sequencing (Immunoseq).
Secondary Endpoint-PD-L1 expression comparison within the Tumor Microenvironment | 1 year for all 4 cohorts to enroll and undergo treatment.
  Identify PD-L1 expression on tumor cells and compare the pretreatment endoscopic biopsies, post-treatment surgical specimens, and historical controls level of PD-L1 expression.
Secondary Endpoint-CD4+ and regulatory T cells expression comparison within the Tumor Microenvironment | 1 year for all 4 cohorts to enroll and undergo treatment.
  Identify CD4+ and regulator T cell infiltration into the tumor microenvironment and compare CD4+ and regulatory T Cell quantity between the pretreatment endoscopic biopsies, post-treatment surgical specimens, and the historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: George Peoples, MD, FACS, Principal Investigator — LumaBridge
Locations (1):
- Clinical Associates of Research Therapeutics of America, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No